CLINICAL TRIAL: NCT06998693
Title: A Single-Center Observational Study on the Impact of Symptom Assessment Timing on the Short-Term Efficacy of 5-ASA Therapy in Patients With Initial-Onset or Relapsed Mild-to-Moderate Active Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Jie Liang, Professor, Xijing Hospital of Digestive Diseases
Other Study IDs: KY20232344-F-1
Record Dates: First submitted 2025-05-06; First posted 2025-05-31 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Ul
Keywords: Ulcerative colitis; 5-aminosalicylic acid; Symptom Assessment Timing; Observational Study
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 4-week Evaluation of Disease Progression: UC patients with initial onset or recurrence whose assessment time interval is set at 4 weeks
  Interventions: Drug: 5-ASA (5-Aminosalicylate); Procedure: Colon Endoscopy Procedure; Diagnostic Test: Blood Routine Test at 4-week; Diagnostic Test: Stool Routine Test at 4-week; Diagnostic Test: Erythrocyte Sedimentation Rate Test at 4-week; Diagnostic Test: C-reactive Protein Test at 4-week; Diagnostic Test: Liver Function Test at 4-week; Diagnostic Test: Kidney Function Test at 4-week
- 8-week Evaluation of Disease Progression: UC patients with initial onset or recurrence whose assessment time interval is set at 8 weeks
  Interventions: Drug: 5-ASA (5-Aminosalicylate); Procedure: Colon Endoscopy Procedure; Diagnostic Test: Blood Routine Test at 8-week; Diagnostic Test: Stool Routine Test at 8-week; Diagnostic Test: Erythrocyte Sedimentation Rate Test at 8-week; Diagnostic Test: C-reactive Protein Test at 8-week; Diagnostic Test: Liver Function Test at 8-week; Diagnostic Test: Kidney Function Test at 8-week
- 12-week Evaluation of Disease Progression: UC patients with initial onset or recurrence whose assessment time interval is set at 12 weeks
  Interventions: Drug: 5-ASA (5-Aminosalicylate); Procedure: Colon Endoscopy Procedure; Diagnostic Test: Blood Routine Test at 12-week; Diagnostic Test: Stool Routine Test at 12-week; Diagnostic Test: Erythrocyte Sedimentation Rate Test at 12-week; Diagnostic Test: C-reactive Protein Test at 12-week; Diagnostic Test: Liver Function Test at 12-week; Diagnostic Test: Kidney Function Test at 12-week

INTERVENTIONS:
Drug: 5-ASA (5-Aminosalicylate) — Specialist doctors decide the administration method of 5-ASA based on the patient's condition (all groups), mainly including topical therapy, or oral therapy (2-4 gram/day).
Procedure: Colon Endoscopy Procedure — Participants in all groups will receive a standard Colon Endoscopy Procedure at 48-week.
Diagnostic Test: Blood Routine Test at 4-week — Participants in will receive a standard Blood Routine Test at 4-week.
  Groups: 4-week Evaluation of Disease Progression
Diagnostic Test: Blood Routine Test at 8-week — Participants in will receive a standard Blood Routine Test at 8-week.
  Groups: 8-week Evaluation of Disease Progression
Diagnostic Test: Blood Routine Test at 12-week — Participants in will receive a standard Blood Routine Test at 12-week.
  Groups: 12-week Evaluation of Disease Progression
Diagnostic Test: Stool Routine Test at 4-week — Participants in will receive a standard Stool Routine Test at 4-week.
  Groups: 4-week Evaluation of Disease Progression
Diagnostic Test: Stool Routine Test at 8-week — Participants in will receive a standard Stool Routine Test at 8-week.
  Groups: 8-week Evaluation of Disease Progression
Diagnostic Test: Stool Routine Test at 12-week — Participants in will receive a standard Stool Routine Test at 12-week.
  Groups: 12-week Evaluation of Disease Progression
Diagnostic Test: Erythrocyte Sedimentation Rate Test at 4-week — Participants in will receive a standard Erythrocyte Sedimentation Rate Test at 4-week.
  Groups: 4-week Evaluation of Disease Progression
Diagnostic Test: Erythrocyte Sedimentation Rate Test at 8-week — Participants in will receive a standard Erythrocyte Sedimentation Rate Test at 8-week.
  Groups: 8-week Evaluation of Disease Progression
Diagnostic Test: Erythrocyte Sedimentation Rate Test at 12-week — Participants in will receive a standard Erythrocyte Sedimentation Rate Test at 12-week.
  Groups: 12-week Evaluation of Disease Progression
Diagnostic Test: C-reactive Protein Test at 4-week — Participants in will receive a standard C-reactive Protein Test at 4-week.
  Groups: 4-week Evaluation of Disease Progression
Diagnostic Test: C-reactive Protein Test at 8-week — Participants in will receive a standard C-reactive Protein Test at 8-week.
  Groups: 8-week Evaluation of Disease Progression
Diagnostic Test: C-reactive Protein Test at 12-week — Participants in will receive a standard C-reactive Protein Test at 12-week.
  Groups: 12-week Evaluation of Disease Progression
Diagnostic Test: Liver Function Test at 4-week — Participants in will receive a standard Liver Function Test at 4-week.
  Groups: 4-week Evaluation of Disease Progression
Diagnostic Test: Liver Function Test at 8-week — Participants in will receive a standard Liver Function Test at 8-week.
  Groups: 8-week Evaluation of Disease Progression
Diagnostic Test: Liver Function Test at 12-week — Participants in will receive a standard Liver Function Test at 12-week.
  Groups: 12-week Evaluation of Disease Progression
Diagnostic Test: Kidney Function Test at 4-week — Participants in will receive a standard Kidney Function Test at 4-week.
  Groups: 4-week Evaluation of Disease Progression
Diagnostic Test: Kidney Function Test at 8-week — Participants in will receive a standard Kidney Function Test at 8-week.
  Groups: 8-week Evaluation of Disease Progression
Diagnostic Test: Kidney Function Test at 12-week — Participants in will receive a standard Kidney Function Test at 12-week.
  Groups: 12-week Evaluation of Disease Progression

SUMMARY:
This study aims to collect the relevant clinical examination results of patients during the 5-ASA treatment period through opportunistic sampling of patients with mild to moderate active ulcerative colitis (UC). The study compares the impact of the time nodes of the first assessment (4th, 8th, and 12th weeks) on the short-term efficacy of 5-ASA. By integrating the dynamic changes of symptom scores and related biomarkers, the study clarifies the time trajectory of symptom relief in patients with mild to moderate UC, identifies the characteristics of early responders and non-responders, and further explores the association between baseline clinical features and treatment responses, thereby assisting in individualized treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

1. According to the diagnostic criteria of the China's 2023 Consensus Opinion on the Diagnosis and Treatment of Inflammatory Bowel Disease, the disease status is newly diagnosed ulcerative colitis (UC) or mild to moderate active UC with remission followed by recurrence (modified Mayo score 3-10 points);
2. Age: 18-59 years old;
3. The attending physician will propose an oral mesalazine or an oral w/ topical mesalazine combined treatment plan based on the patient's condition;
4. Patients who are abble to and are willing to comply with the research protocol can provide a signed and dated written informed consent form.

Exclusion Criteria:

1. Use any form of hormone within the past 14 days;
2. Have received immunosuppressive therapy within the past 90 days;
3. Have used infliximab, adalimumab, or vedolizumab within the past 60 days;
4. Have taken anti-diarrheal drugs within the past 3 days;
5. Have participated in any clinical trial within the past 3 months;
6. Allergic to mesalazine or salicylic acid preparations (except sulfasalazine), including severe adverse reactions, liver and kidney diseases, heart and lung diseases, malignant tumors, etc.;
7. Have had severe liver and kidney diseases, heart and lung diseases, hematological diseases and pancreatic diseases in the past;
8. Pregnant or lactating women;
9. Patients who have withdrawn their informed consent.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study aims to compare the impact of the time point of the first assessment of patients (4th, 8th, and 12th weeks) on the short-term efficacy of 5-ASA on ulcerative colitis. The patients are divided into three groups: the 4-week assessment group, the 8-week assessment group, and the 12-week assessment group, with 60 patients in each group, totaling 180 patients.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
The Endoscopic Remission Rate | 48 weeks From Enrollment
  The primary outcome measure is the endoscopic remission rate at 48 weeks from enrollment, defined as the proportion of patients achieving a Mayo endoscopic subscore of 0 or 1. Participants are adults (18-59 years) with newly diagnosed or relapsing mild-to-moderate ulcerative colitis (modified Mayo score 3-10) receiving oral or oral-plus-topical mesalazine therapy. Patients with recent use of corticosteroids, immunosuppressants, biologics, or other confounding treatments are excluded. Endoscopic assessment is performed at week 48 to evaluate mucosal healing, and the remission rate is calculated based on the number of patients meeting the endoscopic criteria.

SECONDARY OUTCOMES:
The symptom improvement at 12-week after enrollment | 12-week after enrollment
  This outcome measure is symptom improvement at 12 weeks after enrollment, assessed by the change in modified Mayo score from baseline. This score evaluates key ulcerative colitis symptoms, including stool frequency, rectal bleeding, and urgency, with higher scores indicating greater severity. Participants are adults with newly diagnosed or relapsing mild-to-moderate UC receiving mesalazine therapy. Symptom severity is recorded at baseline and at week 12, and improvement is defined as a reduction in the total modified Mayo score, reflecting clinical response to treatment during the 12-week period.
The symptom remission at 12-week after enrollment | 12-week after enrollment
  This outcome measures the symptom remission at 12 weeks post-enrollment in the study population of adult UC patients treated with mesalazine therapy. Eligible participants are those meeting the 2023 Chinese Consensus diagnostic criteria for newly diagnosed or mild-to-moderate active ulcerative colitis (baseline modified Mayo score 3-10), with no recent use of corticosteroids, immunosuppressants, biologics, or anti-diarrheal medications, and without serious comorbidities, concurrent trial participation, or pregnancy. Symptom remission is defined as normal stool frequency and no rectal bleeding or urgency, at the 12-week follow-up visit. This stringent definition indicates minimal disease activity across all symptom domains and is used to evaluate the efficacy of mesalazine in inducing clinical remission by the 12-week mark.
The clinical improvement at 12-week after enrollment | 12-week after enrollment
  This outcome measures the proportion of patients achieving clinical improvement at the 12-week follow-up after enrollment. Clinical improvement is defined as a marked reduction in ulcerative colitis disease activity from baseline. Specifically, a patient must exhibit a decrease in the total modified Mayo score by at least 3 points and at least 30% relative to their baseline score, indicating a significant overall improvement in symptoms. In addition, there must be an improvement in rectal bleeding, evidenced by a decrease of at least 1 point in the rectal bleeding subscore. All participants will be assessed at week 12 post-enrollment to determine if they meet these criteria, reflecting meaningful clinical improvement after 12 weeks of mesalazine therapy.
The clinical remission at 12-week after enrollment | 12-week after enrollment
  Clinical remission at 12 weeks after enrollment is a key secondary outcome measure, defined as achieving a total modified Mayo score of ≤2 with no individual subscore greater than 1 at the 12-week follow-up. This outcome evaluates the effectiveness of 12-week mesalazine therapy (oral or oral-plus-topical) in inducing remission in adult ulcerative colitis patients. Participants are aged 18-59 years and meet the 2023 Chinese Consensus diagnostic criteria for newly diagnosed or mild-to-moderate active UC, with a baseline modified Mayo score between 3 and 10. Patients with recent use of corticosteroids, immunosuppressants, biologic therapies, or anti-diarrheal medications, as well as those in other clinical trials or with serious comorbidities or pregnancy, are excluded. The proportion of patients meeting the clinical remission criteria at week 12 will be determined, providing a clear measure of therapeutic success in this population.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bressler B, Marshall JK, Bernstein CN, Bitton A, Jones J, Leontiadis GI, Panaccione R, Steinhart AH, Tse F, Feagan B; Toronto Ulcerative Colitis Consensus Group. Clinical practice guidelines for the medical management of nonhospitalized ulcerative colitis: the Toronto consensus. Gastroenterology. 2015 May;148(5):1035-1058.e3. doi: 10.1053/j.gastro.2015.03.001. Epub 2015 Mar 4. PMID 25747596
- [Background] Orchard TR, van der Geest SA, Travis SP. Randomised clinical trial: early assessment after 2 weeks of high-dose mesalazine for moderately active ulcerative colitis - new light on a familiar question. Aliment Pharmacol Ther. 2011 May;33(9):1028-35. doi: 10.1111/j.1365-2036.2011.04620.x. Epub 2011 Mar 8. PMID 21385195
- [Background] Hanauer SB, Sandborn WJ, Kornbluth A, Katz S, Safdi M, Woogen S, Regalli G, Yeh C, Smith-Hall N, Ajayi F. Delayed-release oral mesalamine at 4.8 g/day (800 mg tablet) for the treatment of moderately active ulcerative colitis: the ASCEND II trial. Am J Gastroenterol. 2005 Nov;100(11):2478-85. doi: 10.1111/j.1572-0241.2005.00248.x. PMID 16279903
- [Background] Pruitt R, Hanson J, Safdi M, Wruble L, Hardi R, Johanson J, Koval G, Riff D, Winston B, Cross A, Doty P, Johnson LK. Balsalazide is superior to mesalamine in the time to improvement of signs and symptoms of acute mild-to-moderate ulcerative colitis. Am J Gastroenterol. 2002 Dec;97(12):3078-86. doi: 10.1111/j.1572-0241.2002.07103.x. PMID 12492193
- [Background] Levine DS, Riff DS, Pruitt R, Wruble L, Koval G, Sales D, Bell JK, Johnson LK. A randomized, double blind, dose-response comparison of balsalazide (6.75 g), balsalazide (2.25 g), and mesalamine (2.4 g) in the treatment of active, mild-to-moderate ulcerative colitis. Am J Gastroenterol. 2002 Jun;97(6):1398-407. doi: 10.1111/j.1572-0241.2002.05781.x. PMID 12094857
- [Background] Xu L, He B, Sun Y, Li J, Shen P, Hu L, Liu G, Wang J, Duan L, Zhan S, Wang S. Incidence of Inflammatory Bowel Disease in Urban China: A Nationwide Population-based Study. Clin Gastroenterol Hepatol. 2023 Dec;21(13):3379-3386.e29. doi: 10.1016/j.cgh.2023.08.013. Epub 2023 Sep 1. PMID 37660767
- [Background] Baumgart DC, Carding SR. Inflammatory bowel disease: cause and immunobiology. Lancet. 2007 May 12;369(9573):1627-40. doi: 10.1016/S0140-6736(07)60750-8. PMID 17499605